CLINICAL TRIAL: NCT06152653
Title: The Effects of Positive Airway Pressure on the Mucolytic Effects of NAC
Brief Title: The Effects of Positive Airway Pressure on the Mucolytic Effects of NAC (TEAM)
Acronym: TEAM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-39679; 2R01HL080414-13A1 (NIH)
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Asthma; COPD
Keywords: Asthma; COPD; Mucolytic; Mucus Plug; Positive Pressure; NAC
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — N-monoacetylcystine; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NAC via jet nebulizer (Active Comparator): NAC (trade name: Mucomyst) is manufactured by American Regent. The active drug studied here is 10% NAC coadministered with albuterol and delivered via standard jet nebulizer. Participants will each complete 5 treatment visits over the course of 30 days. Each treatment visit will consist of two treatments separated by 4 hours.
  Interventions: Drug: n-acetylcystine (NAC)+ albuterol
- NAC via AeroEclipse-VersaPAP (Experimental): NAC (trade name: Mucomyst) is manufactured by American Regent. The active drug studied here is 10% NAC coadministered with albuterol and delivered via the AeroEclipse-VersaPAP system. Participants will each complete 5 treatment visits over the course of 30 days. Each treatment visit will consist of two treatments separated by 4 hours.
  Interventions: Drug: n-acetylcystine (NAC)+ albuterol; Device: AeroEclipse-VersaPAP System

INTERVENTIONS:
Drug: n-acetylcystine (NAC)+ albuterol — NAC is a mucolytic drug and Albuterol is a bronchodilator.
  Other Names: Mucomyst; NAC
Device: AeroEclipse-VersaPAP System — The AeroEclipse-VersaPAP System combine continuous positive inspiratory pressure and nebulizer in one system.
  Other Names: VersaPAP System
  Arms: NAC via AeroEclipse-VersaPAP

SUMMARY:
The goal of this clinical trial is to determine if positive pressure during inspiration will improve penetration of aerosolized N-Acetylcysteine (NAC) into airway mucus plugs in the lungs of patients with asthma or Chronic Obstructive Pulmonary Disease (COPD).

The main questions it aims to answer are:

* Does delivery of aerosolized NAC with positive inspiratory pressure have a greater effect on mucus plug burden in the lungs than delivery of NAC without positive pressure.
* Does delivery of aerosolized NAC with positive inspiratory pressure have a greater effect on lung function than delivery of NAC without positive pressure.

Participants will be assigned (in a single blind design) to the NAC via jet nebulizer group or the NAC via AeroEclipse-VersaPAP nebulizer group. Participants will each complete 5 treatment visits over the course of 30 days. Each treatment visit will consist of two treatments of a 10% NAC (3 mL) and 2.5 mg albuterol (0.5mL) inhalation solution separated by 4 hours, via the nebulization method specific to their group.

DETAILED DESCRIPTION:
The optimal method for delivering aerosolized N-acetyl cysteine (NAC, Mucomyst) to the airways for the purpose of lysing mucus plugs is not established. The challenge is to ensure that the NAC aerosol penetrates the mucus plug to lyse it. We hypothesize that increasing the inspiratory pressure during aerosol inhalation will improve mixing of NAC with plugs and increase the chance of lysis within the time that the NAC liquid medication "dwells" in the plugged airway segment. Usual nebulizer systems that generate aerosols for inhalation do not allow for application of pressure during inspiration, but the VersaPAP system (from Monaghan Medical Corporation) has this capability. Specifically, the VersaPAP system combines continuous positive pressure during inspiration while the patient inhales aerosol medication, and the pressure will generate viscous fingers in the mucus plugs to aid lysis.

Recent published work from the Fahy lab has revealed that airway mucus plugs can be identified on low dose CT scans of the lungs and quantified using a bronchopulmonary segment based system to generate a measure that quantifies the mucus plug burden in the lung. This CT based mucus plug scoring system provides a predictive and monitoring biomarker for mucus plug pathology in the lungs of patients with asthma and COPD.

This is a single-blind phase 4 clinical trial designed to help determine the optimal method of delivery of aerosolized NAC to patients with mucus-associated lung disease (asthma and COPD). Subjects will be screened for evidence of mucus in their lungs as determined by CT imaging. Eligible participants will then be assigned to the NAC via jet nebulizer group or the NAC via AeroEclipse-VersaPAP nebulizer group and complete 5 treatment visits over the course of 30 days. Each treatment visit will consist of two treatments of a 10% NAC (3 mL) and 2.5 mg albuterol (0.5mL) inhalation solution separated by 4 hours, via the nebulization method specific to their group.

ELIGIBILITY:
Inclusion Criteria:

Asthma Group:

1. Male or female between the ages of 18 to 85 at Visit 1
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
3. Able to perform reproducible spirometry according to American Thoracic Society (ATS) criteria
4. Clinical history of asthma per patient report or medical record
5. Asthma requiring treatment with inhaled corticosteroids (ICS) or biologic therapy for 3 months or greater
6. Computed Tomography (CT) mucus score ≥ 3 (done as part of screening)
7. There is no lower threshold on Forced Expiratory Volume in the first second (FEV1), which means the study will attempt to enroll all patients regardless of asthma severity. However, eligible participants will need to demonstrate ability to tolerate study treatment reflected by a post-treatment FEV1 ≥ 80% of pre- treatment, pre-bronchodilator FEV1. Participants who have a >20% drop in FEV1 after receiving any study treatment will be excluded from the study.
8. For participants with known mucus plugging on CT: no limit on FEV1;

For participants with unknown mucus plugging: FEV1<70% predicted

COPD Group:

1. Males or females between the ages 18 to 85 at the time of visit 1.
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
3. History of COPD per patient report or medical record and confirmed by an FEV1/FVC ratio of under 70%.
4. Current or former smoker with a history of at least 10 pack-years of smoking.
5. CT mucus score ≥ 3
6. There is no lower threshold on FEV1, which means the study will attempt to enroll all patients regardless of COPD severity. However, eligible participants will need to demonstrate ability to tolerate study treatment reflected by a post-treatment FEV1 ≥ 80% of pre- treatment, pre-bronchodilator FEV1. Participants who have a >20% drop in FEV1 after receiving any study treatment will be excluded from the study.
7. For participants with known mucus plugging on CT: no limit on FEV1; For participants with unknown mucus plugging: FEV1<50% predicted

Exclusion Criteria:

1. A history of medical disease, which in the opinion of the investigator may put the subject at extra risk from study-related procedures or because the disease may influence the results of the study.
2. Currently pregnant
3. URI in past 10 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in mucus plug score | 1 week before treatment to 1 week post treatment, an average of 6 weeks
  The primary outcome is the % change in mucus plug score from 1 week before treatment to 1 week post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, MS, Principal Investigator — Professor of Medicine
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hays SR, Fahy JV. The role of mucus in fatal asthma. Am J Med. 2003 Jul;115(1):68-9. doi: 10.1016/s0002-9343(03)00260-2. No abstract available. PMID 12867239
- [Background] DUNNILL MS. The pathology of asthma, with special reference to changes in the bronchial mucosa. J Clin Pathol. 1960 Jan;13(1):27-33. doi: 10.1136/jcp.13.1.27. PMID 13818688
- [Background] Chui JY, de Anna P, Juanes R. Interface evolution during radial miscible viscous fingering. Phys Rev E Stat Nonlin Soft Matter Phys. 2015 Oct;92(4):041003. doi: 10.1103/PhysRevE.92.041003. Epub 2015 Oct 28. PMID 26565159
- [Background] Tang M, Elicker BM, Henry T, Gierada DS, Schiebler ML, Huang BK, Peters MC, Castro M, Hoffman EA, Fain SB, Ash SY, Choi J, Hall C, Phillips BR, Mauger DT, Denlinger LC, Jarjour NN, Israel E, Phipatanakul W, Levy BD, Wenzel SE, Bleecker ER, Woodruff PG, Fahy JV, Dunican EM. Mucus Plugs Persist in Asthma, and Changes in Mucus Plugs Associate with Changes in Airflow over Time. Am J Respir Crit Care Med. 2022 May 1;205(9):1036-1045. doi: 10.1164/rccm.202110-2265OC. PMID 35104436